CLINICAL TRIAL: NCT05783193
Title: TGIR (Traditional Gastrointestinal Remedy) Randomized Placebo-controlled Healthy Subject Study
Brief Title: TGIR Randomized Placebo-controlled Healthy Subject Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Resilience Biosciences Inc (RBI) (Unknown)
Responsible Party: Principal Investigator, Pouya Azar, Medical Manager, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H21-03899
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover trial with healthy volunteers to delineate additional information on a Health Canada-approved natural health product.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TGIR (Traditional Gastrointestinal Remedy) (Experimental): TGIR (500mg/capsule), 1.0g (2 capsules)
  Interventions: Drug: TGIR (Traditional Gastrointestinal Remedy)
- Control (Microcrystalline cellulose) (Placebo Comparator): Placebo control (2 capsules)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TGIR (Traditional Gastrointestinal Remedy) — TGIR botanical formulation
  Arms: TGIR (Traditional Gastrointestinal Remedy)
Drug: Placebo — Placebo capsules
  Arms: Control (Microcrystalline cellulose)

SUMMARY:
The primary research objective of this study is to confirm the absence of side-effects and explore any analgesic properties of the botanical formulation TGIR (Traditional Gastrointestinal Remedy) in healthy participants.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, crossover, clinical trial with 24 healthy volunteers. Participants will be randomized to receive each of the two treatments, TGIR (500mg/capsule, total 1.0g) followed by Placebo (2 matching capsules), or vice-versa, with a week between treatments. Participants will remain in the clinic for a 4-hr observation period each day for a total of 2 clinic visits. During the course of treatment, participants will receive physiological monitoring: heart rate and blood pressure. Any adverse events and side effects will be documented throughout the study, in addition to participant feedback and perceived effects. On each day of treatment (TGIR and placebo-control), participants will receive a standardized test of analgesia using Brief Thermal Sensitization (BTS) and measures of reaction time using a computer-based Psychomotor Vigilance Task (PVT).

ELIGIBILITY:
Inclusion Criteria:

* Self-reported to be in good health
* Between the ages of 18 and 65
* No chronic pain diagnosis
* Willing and able to follow study protocol and schedule

Exclusion Criteria:

* Participants who are pregnant, breastfeeding or planning to become pregnant during the course of the study
* History or current clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, neurological, or psychiatric disease that may pose a significant safety risk or diminish a participant's ability to undergo all study procedures and assessments
* Participants who have been diagnosed with a severe medical or psychiatric condition
* Participants who are actively taking pain medication in the past 7 days
* COVID-19 positive and/or showing symptoms of COVID-19
* Concurrent use of other supplements containing sedative types of herbs, such as valerian, skullcap, hops, california poppy, passiflora, and cannabis during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Standardized heat sensitivity testing - Brief Thermal Sensitization (BTS) | 30-60min post-treatment
  Participants rate the painfulness of the heat stimulation on a paper 100 mm Visual Analogue Scale anchored with the descriptors "no pain" (0 mm) and "worst pain imaginable" (100 mm).
Measure of reaction time - Psychomotor vigilance task (PVT) | 60min post-treatment
  PVT performance on a computer-based test measures lapses, defined as reaction times exceeding 500 msec or failure to react.

SECONDARY OUTCOMES:
Physiological monitoring - Heart rate | Recording every 30min over 4 hours post-treatment
  Heart rate monitoring
Physiological monitoring - Blood pressure | Recording every 30min over 4 hours post-treatment
  Blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Pouya Rezazadeh-Azar, MD, Principal Investigator — University of British Columbia
Locations (1):
- Joseph & Rosalie Segal & Family Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No